CLINICAL TRIAL: NCT05487469
Title: Thymosin α1 Use in Rheumatic Heart Disease Patients Undergoing Cardiac Surgery on Cardiopulmonary Bypass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Principal Investigator of Cardiovascular Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5A Plan IV
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Rheumatic Heart Disease; Cardiopulmonary Bypass; Immunotherapy
MeSH Terms: conditions — Rheumatic Heart Disease | interventions — Thymalfasin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thymosin alpha 1 (Experimental)
  Interventions: Drug: Thymosin Alpha1
- Blank control (Sham Comparator)
  Interventions: Other: Blank Control

INTERVENTIONS:
Drug: Thymosin Alpha1 — Thymosin alpha 1, 1.6mg injection hypodermic (I.H), every 12 hours for 5 days at least during the ICU admission. The administration will be terminated any day during the treatment when the patient is deemed as qualified for ICU discharge or dead
  Arms: Thymosin alpha 1
Other: Blank Control — the Control group did not receive Thymosin alpha 1 or any placebo.
  Arms: Blank control

SUMMARY:
Rheumatic heart disease usually accompanied by weakened immune function. And the cardiopulmonary bypass further aggravating the decline of immune function. Therefore, the prevention of Postoperative immune function collapse is of great clinical value, and immunomodulatory therapy with thymosin alpha

1 may be beneficial. This study was designed to test the hypothesis that the administration of thymosin alpha 1 will Improve the immune function and prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients are conformed to 2004 WHO guidelines for Rheumatic fever and rheumatic heart disease;
* Patients planning to undergo cardiac surgery were enrolled.
* The patients' age between 18 ~80 years old.
* Agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Patients allergic to Thymosin α1;
* Lactating women and pregnant women;
* Patients with mental diseases, drug and alcohol dependence;
* Refuse to participate in this study and refuse to sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The highest Sequential Organ Failure Assessment (SOFA) score of 5 days after surgery | 5 days after surgery

SECONDARY OUTCOMES:
30-day mortality | 30 days after randomization
  Death from any cause of 30 days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of nanjing medical university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided